CLINICAL TRIAL: NCT01038128
Title: Antiglutamatergic Treatment of Bulimia Nervosa and Body Dysmorphic Disorder: An Open-Label Trial of Memantine
Brief Title: An Open Label Trial of Memantine in the Treatment of Bulimia Nervosa and Body Dysmorphic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, James I. Hudson, MD, Professor of Psychiatry, Harvard Medical School, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-P-001901
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Results first posted 2012-06-12 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Bulimia Nervosa; Body Dysmorphic Disorder
Keywords: Bulimia nervosa; Bulimia; Body dysmorphic disorder; Eating disorders; Body image; Binge eating; purging
MeSH Terms: conditions — Bulimia Nervosa; Body Dysmorphic Disorders; Bulimia; Feeding and Eating Disorders | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Memantine (Experimental): Memantine, 10-40 mg daily
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine — Drug: Memantine, 10-40 mg daily
  Other Names: Namenda

SUMMARY:
The primary objective of this 13-week clinical trial is to test the hypothesis that treatment with Memantine will significantly improve the symptoms of those suffering from either bulimia nervosa, purging type or suffering from body dysmorphic disorder.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to test the hypothesis that treatment with Memantine, an anti-glutamatergic drug, will significantly improve the core symptoms of those suffering from either bulimia nervosa, purging type or suffering from body dysmorphic disorder.

We will test this hypothesis by performing a 13-week open label study investigating the use of memantine, at a dose of 10-40mg daily, as a treatment for patients with either bulimia nervosa or body dysmorphic disorder. Improvement for patients with bulimia nervosa will be assessed using the Frequency of binge eating and vomiting as recorded in diary card, Eating Disorder Evaluation (EDE), and the Yale-Brown-Cornell Eating Disorders Scale (YBC-EDS). Improvement for patients with body dysmorphic disorder will be assessed using the the Yale-Brown-Cornell Eating Disorders Scale (YBC-EDS) and Brown Assessments of Beliefs Scale. In addition both groups will also receive the Clinical Global Impression (CGI) Severity and Improvement Scales (clinician rated), Patient Global Impression of Improvement (PGI-Improvement), Montgomery Asberg Depression Rating Scale (MADRS), Hamilton Anxiety Rating Scale (HAM-A), Barratt Impulsiveness Scale (BIS), Version 11, Sheehan Disability Scale (SDS), and Columbia Suicide Severity Rating Scale (C-SSRS).

ELIGIBILITY:
Inclusion Criteria: Bulimia Nervosa

* Participants must meet DSM-IV criteria for a current diagnosis of bulimia nervosa as determined by the Structured Clinical Interview for DSM-IV (SCID) and Eating Disorder Examination (EDE).
* Participants must report an average of 3 or more binges and vomiting episodes per week in the 2-week period prior to the screening visit.
* Male or Female between 18 and 65 years of age, inclusive.
* Female participants must be: postmenopausal for at least one year, surgically sterile, or practicing an effective method of birth control (e.g., prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization, abstinence and agreeing to continue abstinence or to use one of the acceptable methods of contraception just enumerated should sexual activity commence) before entry and throughout the study; and have a negative serum pregnancy test at the screening visit.
* Participants must have observed a designated washout period of at least seven days or a period equal to five half-lives of prohibited medications.
* Participants must be able to take oral medication, adhere to the medication regimens, and be willing to return for regular visits.
* Participants must be able and willing to read and comprehend written instructions and comprehend and complete all scales and questionnaires required by the protocol.
* Participants must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Inclusion Criteria: Body Dysmorphic Disorder

Inclusion criteria for participants with body dysmorphic disorder are identical to those for bulimia nervosa above, with the following differences in the first two criteria:

* Participants must meet DSM-IV criteria for a current diagnosis of body dysmorphic disorder as determined by the SCID.
* Participants must exhibit a score of ≥ 20 on the Body Dysmorphic Disorder Version of the Yale Brown Obsessive Compulsive Scale (BDD-YBOCS) at a score of ≥ 5 on the first three items of the BDD-YBOCS, which are the items that assess the DSM-IV criteria for Body Dysmorphic Disorder.

Exclusion Criteria for both Bulimia Nervosa and Body Dysmorphic Disorder:

* Participants with a lifetime diagnosis of schizophrenia, other psychotic disorder, or bipolar disorder as defined by DSM-IV and supported by the SCID.
* Participants with clinically significant current depression or who, in the investigators' judgment, might require intervention with either pharmacological or non-pharmacological therapy for major depressive disorder over the course of the study.
* Participants judged clinically to be at suicidal or homicidal risk by the study physician.
* Participants meeting DSM-IV criteria for any form of substance dependence or abuse (with the exception of nicotine or caffeine dependence) within 3 months prior to the screening visit.
* Participants meeting DSM-IV criteria for anorexia nervosa within 3 months prior to the screening visit.
* Participants with a current DSM-IV diagnosis of an organic mental disorder.
* Participants who have begun to receive formal psychotherapy (cognitive-behavioral therapy, interpersonal therapy or self-guided cognitive-behavioral therapy) for bulimia nervosa within 6 months prior to the screening visit.
* Participants who display a positive urine screen for drugs of abuse (phencyclidine, cocaine, amphetamines, tetrahydrocannabinol, and opiates) at the screening visit.
* Participants who have previously received memantine for any reason.
* Participants who have received an investigational medication within 30 days of the screening visit.
* Participants who are pregnant or lactating.
* Participants with a body mass index (BMI) less than 18.5 or greater than 35.
* Participants who have abused ipecac as a method of purging within the past 2 years.
* Participants who exhibit a serum potassium level of less than 3.0 mEq/L.
* Participants with thyroid-stimulating hormone concentrations outside the range of 0.5-5.0 lU/mL.
* Participants with clinically significant or unstable medical conditions
* Participants who in the opinion of the investigator should not be enrolled in the study because of the precautions, warnings or contraindications sections of the prescribing information for memantine
* Employees of the investigator, individuals with direct involvement in studies under the direction of the study investigators, as well as family members of the employees of the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James I Hudson, M.D., Sc.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Memantine
Started | 5
Baseline Visit | 3
Completed | 1
Not Completed | 4
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Memantine
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (18.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Binge Eating and Self-induced Vomiting Episodes
Description: Number of self-reported binge eating and self-induced vomiting episodes during the week prior to the Baseline and Endpoint Visits.
Time Frame: Baseline to 12 weeks
Population: One subject completed. The remaining two subjects' last observation was carried forward.
Measure: Mean (Standard Deviation); unit: number of episodes
Groups:
- Memantine: Number of Binge Eating and Purging Episodes at Baseline and Endpoint
Arm/Group | Memantine
Number analyzed (Participants) | 3
number of episodes
  Binge Eating Baseline | 20.67 (14.74)
  Binge Eating Endpoint | 31.33 (35.25)
  Purging Baseline | 21.67 (27.30)
  Purging Endpoint | 36.67 (54.93)

2. Primary Outcome: Ratings of Eating Pathology
Description: Ratings obtained from the self-induced vomiting and laxative misuse sections of the Eating Disorder Examination. The scale asks participants to calculate discreet episodes of self-induced vomiting and laxative misuses over the period of four weeks. Generally, the value obtained is the number of occurrences. However, in cases where the number of occurrences was too great to be calculated, the number "777" was used. The scale is therefore open-ended, with higher numbers coinciding with a greater number of episodes.
Time Frame: Baseline to 12 weeks
Population: One subject completed. The remaining two subjects' last observation was carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Memantine: Ratings at Baseline and Endpoint
Arm/Group | Memantine
Number analyzed (Participants) | 3
units on a scale
  Baseline Data | 101.33 (71.07)
  Endpoint Data | 38.67 (30.27)

3. Primary Outcome: Clinical Global Impression Scale
Description: Disorder severity is measured based on the Clinical Global Impression Scale. The scale ranges from 1 unit (Not at all ill) to 7 units (extremely ill).
Time Frame: Baseline to 12 weeks
Population: One subject completed. The remaining two subjects' last observation was carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 3
units on a scale
  Baseline Data | 5 (0)
  Endpoint Data | 4 (1.41)

4. Primary Outcome: Body Dysmorphic Disorder Version of the Yale Brown Obsessive Compulsive Scale
Description: The scale ranges from 0 to 91 units, with 0 representing the least ill and 91 representing the most ill.
Time Frame: Baseline to 12 weeks
Population: One subject completed. The remaining two subjects' last observation was carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Memantine
Number analyzed (Participants) | 3
units on a scale
  Baseline Data | 57.67 (0.58)
  Endpoint Data | 48.67 (6.51)

5. Primary Outcome: Brown Assessments of Belief Scale
Description: The range for this scale is 0 to 28 units, with 0 representing the least ill and 28 representing the most ill.
Time Frame: Baseline to 12 weeks
Population: This scale was only administered to participants with Body Dysmorphic Disorder. No participants with BDD completed the Baseline Visit and, therefore, no results were available to analyze.
Groups:
- Baseline Data: Ratings at Baseline and Endpoint.
Arm/Group | Baseline Data
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Memantine
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=3)
Constipation (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Pain when closing eyes (Eye disorders) | 1 (1)
Constant eye pressure (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No